CLINICAL TRIAL: NCT02733770
Title: Comparison in Portal Flow After Sleeve Gastrectomy and Mini Gastric Bypass
Brief Title: Chances in Portal System Flow After Two Bariatric Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Sergio Gabriel Susmallian, Head of the Dpartment of Surgery, Assuta Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AMC0416
Record Dates: First submitted 2016-03-26; First posted 2016-04-12 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Portal Vein Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleeve gastrectomy (Active Comparator): US DOopler for Patient with BMI of 40 or more than 35 with co-morbidities underwent Sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy; Procedure: Laparoscopic mini gastric bypass
- Mini Gastric Bypass (Active Comparator): US DOopler for Patient with BMI of 40 or more than 35 wtih co-morbidities underwent mini gastric bypass
  Interventions: Procedure: Laparoscopic sleeve gastrectomy; Procedure: Laparoscopic mini gastric bypass

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Doppler ultrasound.
Procedure: Laparoscopic mini gastric bypass — Doppler ultrasound.

SUMMARY:
Obesity if a health endemic problem over the entire world. Bariatric surgery is the best chance for those patients with morbid obesity to loss weight and to maintain the loosed weight.

Metabolic surgery is the new name for bariatric surgery like sleeve gastrectomy and gastric by pass due to the recognized changes in the homeostasis of the hormonal secretion responsive to the hunger status. After sleeve gastrectomy we observe many patients with thrombus of the portal vein system. This phenomena may be attributed to changes in the portal flow due to devascularization of the great curvature of the stomach.

The aim of the study is to compare the portal flow by intra-operative Doppler ultrasound before and after surgery of the two procedures as sleeve gastrectomy and gastric bypass, were the vascularization is not changed by the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for bariatric surgery for the bariatric surgery committee.
* Primary procedure
* No hypercoagulability status know

Exclusion Criteria:

* Hypercoagulability status
* patients after any abdominal surgery of the forgut

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Measurement of Portal flow | three month
  physiological parameter

SECONDARY OUTCOMES:
Determine the relation between the operation and thrombosis | three month
  physiological parameter and number of thrombosis found. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta MC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No